CLINICAL TRIAL: NCT07279272
Title: The Effect of the Human Regenerator Jet Device on the Quality of Life of Adult Individuals [HR-QoL]
Acronym: HR-QoL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Athens (Other)
Collaborators: THE ENDOCRINE UNIT OF THE UNIVERSITY OF ATHENS (Unknown)
Responsible Party: Principal Investigator, Eumorphia Remboutsika, Researcher B ( Associate Professor Level), University Research Institute for the Study of Genetic & Malignant Disorders in Childhood
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: RPURI9023; License 62101 (Other: EuroQoL)
Record Dates: First submitted 2025-11-18; First posted 2025-12-12 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Chronic Stress; Chronic Fatigue; Chronic Pain; Post-COVID / Long-COVID
Keywords: Cold Atmospheric Plasma; Human Regenerator Jet; Human Regenerator Power Jet; Human Regenerator Sports Jet; Human Regenerator Med Jet; Human Regenerator
MeSH Terms: conditions — Chronic Pain; Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Intervention Model Description: HR-QoL single-blind crossover study evaluates the effects of a novel cold atmospheric plasma jet producing device, the Human Regenerator Power Jet device (HR) (System4 Technologies GmbH, Germany) for individuals who suffer from chronic stress, chronic pain, chronic fatigue syndrome, sleep disorders, and Post-COVID/Long-COVID Syndrome, all conditions that affect the QoL among adults worldwide. The HR-QoL study has solicited 40 participants randomized into two groups (A & B). Group A (20 adults) was treated at the HR under CAP conditions (CAP Effect) (10 sessions), followed by a 1-month wash-out period, before treatment at the HR under AIR Conditions (Sham Device-Placebo Effect). Group B (20 adults) was treated at the HR under AIR conditions (Sham Device-Placebo Effect) followed by a 1-month wash-out period, before treatment at the HR under CAP Conditions (Cap Effect). The participants are not aware whether they are subjected to CAP or AIR from the device.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CAP to AIR (Active Comparator): Group A (20 adults) were subjected to Cold Atmospheric Plasma (10 sessions) generated by the Human Regenerator jet device (Active Device-CAP Effect), followed by a 1-month wash-out period, before being subjected to AIR (10 sessions) (Sham Device-Placebo Effect).
  Interventions: Device: Cold Atmospheric Plasma; Device: Atmospheric Air
- AIR to CAP (Sham Comparator): Group B (20 adults) were subjected to AIR (10 sessions) generated by the Human Regenerator jet device (Sham Device-Placebo Effect) followed by a 1-month wash-out period, before being subjected to Cold Atmospheric Plasma conditions (10 sessions) (Active Device-Cap Effect)..
  Interventions: Device: Cold Atmospheric Plasma; Device: Atmospheric Air

INTERVENTIONS:
Device: Cold Atmospheric Plasma — The Human Regenerator Jet Device CAP Effect interventions include a 30 minute exposure of the subjects, every other day, with Cold Atmospheric Plasma, a total of 10 sessions
Device: Atmospheric Air — The Human Regenerator Jet Device AIR Effect interventions include a 30 minute exposure of the subjects, every other day, to Atmospheric Air, a total of 10 sessions

SUMMARY:
This cross-over single-blinded study aims to evaluate the effect of a novel cold atmospheric plasma jet-producing device, the Human Regenerator Power Jet device, for individuals who suffer from chronic stress, chronic pain, chronic fatigue, sleep disorders, and Post-COVID/Long-COVID Syndrome, all conditions that affect the QoL among adults in Greece and worldwide.

DETAILED DESCRIPTION:
Introduction: Plasma medicine is a novel, exciting, young interdisciplinary scientific field, emerging from the interaction of physicists, biologists, and medical doctors. Plasma is the fourth matter, often defined as an ionized gas produced by the disintegration of polyatomic gas molecules or the removal of electrons from monatomic gas shells, with the following strict criteria: plasma must be a) macromolecularly neutral (quasi-neutrality); b) Debye shielding; c) frequency. As a result, plasma can be defined as "a quasi-neutral gas containing many interacting free electrons and ionized atoms and molecules, which have collective behavior caused by long-range coulomb forces", and their motion gives rise to electric fields and generates currents and magnetic fields. Plasma is classified into high-temperature, thermal, and non-thermal categories. In high temperature, all particles (both electrons and heavy particles) have the same temperature, and are thus in thermal equilibrium. Non-thermal (non-equilibrium) plasma engulfs particles that are not in thermal equilibrium. This plasma is termed "cold plasma". Cold plasma discharge can be achieved at both low pressure and atmospheric pressure. Low pressure cold plasma was first applied for surface decontamination in a more effective manner than conventional sterilization in the 1960s; by contrast, Cold Atmospheric Plasma (CAP) was applied in 1990s.

CAP is ideal for use in modern medicine because : a) it can be generated easily from a portable device with easier direct access to affected cells and tissues, b) all animal and human tissues contain water and its presence is undesirable in low pressure conditions, c) its ability to reduce microbial load makes it a good option to combat increasing antibiotic resistance, and d) CAP-generating devices have relatively low manufacturing costs. As a result, accessible, efficient, and inexpensive CAP devices can reduce the financial burden imposed on the health budget by conventional treatments.

All plasma devices used in clinical practice are intended to prevent harm to healthy cells. They undergo multistep testing and are associated with no significant side effects. Nevertheless, the proper CAP dosage must be continuously monitored, adjusted for each treatment, with an important parameter to be the distance between the plasma jet source and human skin. Hypothetically speaking, it could not be excluded that CAP does not have some minimal negative effects at the molecular level; these are still subject to ongoing analysis, but results so far suggest that hypothetically unproven adverse effects are outweighed by the enormous benefits of CAP.

Current analyses of CAP effects have concentrated mostly on cells in culture and animal models. Although these efforts are more accessible and easier to conduct, wider testing of CAP effects in disease and regenerative medicine studies in human patients could only be beneficial. Nowadays, CAP is mostly employed in aesthetic procedures; however, its use in more serious medical conditions, such as acute and chronic wounds, oral bacterial infections, and potentially in tumour therapy, is subject to ongoing research. The use of CAP in routine clinical practice in medicine could advance the therapeutic process into a less invasive and distressing process for patients, while also significantly reducing the financial burden of existing treatments in Europe and worldwide.

Aim of the Study: This cross-over single-blinded study evaluates the effect of a novel CAP jet-producing device, the Human Regenerator Power Jet (CE 2022), for individuals who suffer from chronic stress, chronic pain, chronic fatigue, sleep disorders, and Post-COVID/Long-COVID Syndrome, all conditions that affect the QoL among adults in Greece and worldwide [HR-QoL].

Participants: The HR-QoL study has solicited 40 participants randomized into two groups (A & B). Group A (20 adults) was treated at the HR under CAP conditions (CAP Effect) (10 sessions), followed by a 1-month wash-out period, before treatment at the HR under AIR Conditions (Sham Device-Placebo Effect). Group B (20 adults) was treated at the HR under AIR conditions (Sham Device-Placebo Effect) followed by a 1-month wash-out period, before treatment at the HR under CAP Conditions (Cap Effect). The participants were not aware whether they were subjected to CAP or AIR from the device. The HR-QoL study was conducted among adult residents of Greece, according to the World Medical Association Declaration of Helsinki (2013). In the HR-QoL study, "adults" are defined as individuals no younger than 18 years old. The eligible list of participants has been evaluated by the Endocrine Unit of the University of Athens (NKUA).

ELIGIBILITY:
Inclusion Criteria Clinical and laboratory diagnosis of chronic stress/chronic pain/chronic fatigue/Long Covid Criteria:

Exclusion Criteria include:

1. Pregnancy or Breast-feeding period
2. Participation on another Stress related study
3. Patients with implanted devices
4. Patients with major psychiatric disorders
5. Refusal to participate in the study

Ages: 18 Years to 94 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-07-09 (Actual); Primary Completion 2025-07-22 (Actual); Study Completion 2025-07-22 (Actual)

PRIMARY OUTCOMES:
EURO-QOL Quality of Life Health Assessment (License no. 62101) | The time frame ranges from enrollment to completion in 10-11 weeks, with four time points: T1: Enrollment date; T2: 3 weeks; T3: 7 weeks; T4: 10 weeks-Completion date.
  The 5-level EQ-5D version (EQ-5D-5L) was introduced by the EuroQol Group in and it essentially consists of 2 pages: the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS). The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions (1-digit number/dimension), The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state and reflects to the overall health state of each individual (0-1 scale). The EQ VAS records the patient's self-rated health on a vertical visual analogue scale where the endpoints are labelled 'The best health you can image' and 'The worst health you can image' (0-100 scale).

CONTACTS AND LOCATIONS:
Overall Officials: Eumorphia Remboutsika, PhD, Principal Investigator — University Research Institute for the Study of Genetic & Malignant Disorders in Childhood; George P Chrousos, MD, PhD, Study Director — University Research Institute
Locations (1):
- The Endocrine Unit of the University of Athens, Athens, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Human Regenerator Jet Device — https://system4-technologies.com/